CLINICAL TRIAL: NCT04879173
Title: The Clinical Value of Microvascular Ultrasonography in Real-time Differential Diagnosis of Thyrotoxic Patients Between Hyperthyroidism and Thyroiditis
Brief Title: Clinical Value of Microvascular Ultrasonography in Real-time Differential Diagnosis of Thyrotoxic Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Dong Jun Lim (Other)
Responsible Party: Sponsor-Investigator, Dong Jun Lim, professor, Seoul St. Mary's Hospital
Organization: Seoul St. Mary's Hospital (Other)
Other Study IDs: Project name 2
Record Dates: First submitted 2021-05-04; First posted 2021-05-10 (Actual); Last update posted 2021-05-10 (Actual); Status verified 2021-05

CONDITIONS: Hyperthyroidism/Thyrotoxicosis
MeSH Terms: conditions — Hyperthyroidism; Thyrotoxicosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Hyperthyroidism caused by Graves' disease
  Interventions: Device: RS85 Ultrasound device
- Hyperthyroidism caused by painless/subacute thyroiditis
  Interventions: Device: RS85 Ultrasound device

INTERVENTIONS:
Device: RS85 Ultrasound device — RS85 Ultrasound device manufactured by Samsung Medison

SUMMARY:
This study aims to verify the clinical value of thyroid ultrasound with microvascular flow imaging in thyrotoxic patients for differential diagnosis between hyperthyroidism and thyroiditis. We intend to use the RS85 Ultrasound device manufactured by Samsung Medison. Graves' disease and painless thyroiditis/subacute thyroiditis are the main cause of thyrotoxicosis.

Precise discrimination between Graves' disease and painless thyroiditis/subacute thyroiditis is clinically very important in determining treatment methods, such as the prescription of antithyroid drugs. Primary endpoint was to verify the value of vascularity index, defined by Blood pixel in range of image / Total pixel in range of image .Seondary endpoint was to verify the superiority value of Microvascular flow imaging to discriminate thyrotoxicosis patients compared with Color doppler/ Power doppler ultrasound imaging and conventional ultrasound imaging.

DETAILED DESCRIPTION:
Thyrotoxicosis refers to the appearance of various clinical symptoms or signs due to and excessive increase of thyroid hormone in the body. Graves' disease, which causes thyrotoxicosis, is one of the most common autoimmune diseases and is known to account for 0.5% of the population. Precise discrimination between Graves' disease and painless thyroiditis/subacute thyroiditis is clinically very important in determining treatment methods.

The Microvascular flow imaging technology is expected to show higher sensitivity and accuracy than conventional color Doppler images in differentiating patients between Graves' disease and painless thyroiditis/subacute thyroiditis. We enrolled thyrotoxicosis patients in their initial presentation and used RS85 Ultrasound device manufactured by Samsung Medison to discriminate Graves' disease and painless thyroiditis/subacute thyroiditis. Power / Color doppler ultrasound imaging and conventional ultrasound imaging were used. Tranverse and longitudinal plane of the dominant lobe were selected for imaging. Doppler Adler's method was used to asscess vascularization. To assess the vascularity index, which is defined by Blood pixel in range of image / Total pixel in range of image, we selected the total tranverse plane of the thyroid as range of image.

ELIGIBILITY:
Inclusion Criteria:

* Initial presentation with thyrotoxicosis

Exclusion Criteria:

* Past history of thyroidectomy
* Factitious thyrotoxicosis
* Unable for ultrasound

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patient with thyrotoxicosis initially presented at hospital.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2020-10-14 (Actual); Primary Completion 2021-10 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
The optimal value of vascular index for differentiating the thyrotoxicosis reason | 12 months

SECONDARY OUTCOMES:
The superiority value of Microvascular flow imaging | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Dong Jun Lim, MD, PhD, Study Director — the Catholic Univerisity of Korea
Locations (1):
- Seoul St. Mary hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Baek HS, Park JY, Jeong CH, Ha J, Kang MI, Lim DJ. Usefulness of Real-Time Quantitative Microvascular Ultrasonography for Differentiation of Graves' Disease from Destructive Thyroiditis in Thyrotoxic Patients. Endocrinol Metab (Seoul). 2022 Apr;37(2):323-332. doi: 10.3803/EnM.2022.1413. Epub 2022 Apr 13. PMID 35413779